CLINICAL TRIAL: NCT04703959
Title: Glaucoma and Sleep Quality
Acronym: POLY-GLAUCOMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.227; 2020-A01949-30 (Other: ID RCB)
Record Dates: First submitted 2020-12-14; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- glaucomatous subjects (50): Subjects included in the MARS database of CHU Grenoble-Alpes with available polysomnographic data and with the following ophthalmological characteristics:
  * increase in intraocular pressure (IOP before treatment greater than 21 mmHg) with characteristic alterations of the optic nerve (pathological papillary excavation, papillary pallor, papillary atrophy) with corresponding alterations and characteristics of the visual field. The visual field should be considered reliable (European criteria (European Glaucoma Society, 1999).
  * Patients whose age is greater than or equal to 18 years
  * Male or female patients
  * Patients not objecting to the study
  * Affiliation to a social security scheme or beneficiary of such a scheme
  Interventions: Other: polysomnography
- non glaucomatous subjects (100): Subjects included in the MARS database of CHU Grenoble-Alpes with available polysomnographic data and with the following ophthalmological characteristics:
  * no known ophthalmological pathologies, with an ophthalmological examination on telephone examination - in the 2 years preceding the polysomnographic examination - normal apart from minor refractive disorders (myopia with spherical equivalent less than -6 diopters or hyperopia with spherical equivalent less than 3 diopters).
  * Patients whose age is greater than or equal to 18 years
  * Male or female patients
  * Patients not objecting to the study
  * Affiliation to a social security scheme or beneficiary of such a scheme
  Interventions: Other: polysomnography

INTERVENTIONS:
Other: polysomnography — polysomnography is already done for all patients

SUMMARY:
This study is a observational, prospective, case-control, monocentric study.

The main objective is to study the polysomnographic characteristics of sleep in glaucomatous and non-glaucomatous subjects, using data collected in the MARS database of CHU Grenoble-Alpes, to compare the total sleep time of glaucomatous and non-glaucomatous subjects, measured during the polysomnographic examination collected in the database.

The secondary objectives are the exhaustive characterization of the sleep architecture in glaucomatous and non-glaucomatous subjects, from data collected in the MARS database of the CHU Grenoble-Alpes

* Length of sleep period
* Time spent in phase 1, 2, 3 and 4
* Micro-alarm clocks index
* Time with arterial oxygen saturation less than 90%
* Apnea-hypopnea index

DETAILED DESCRIPTION:
Glaucoma is an eye and neurodegenerative disease characterized by progressive destruction of optic nerve cells (retinal ganglion cells), affecting vision but also the retino-hypothalamic pathway leading to the suprachiasmatic nuclei and helping to synchronize nycthemeral rhythms.

It can therefore be suggested that glaucoma may affect the structure and quality of sleep. Few studies on the subjects of sleep quality and architecture have been performed to date, and all are either small series of cases without a comparator group, or studies based on questionnaires but without polysomnographic examination. The results of studies carried out to date are conflicting.

The subject is important because glaucoma is a frequent disease (1 to 1.2 million subjects in France and 75 to 90 million in the world), and could potentially be a frequent cause of disturbance of the quality of sleep.

The CHU Grenoble-Alpes has a large database (MARS Cohort) including polysomnographic examinations of glaucomatous and non-glaucomatous subjects. The objective of this study is to characterize the sleep parameters (sleep time, sleep period, sleep stages, sleep efficiency, cycles per night, micro-arousal index, etc.) in glaucomatous and non-glaucomatous subjects, by controlling any possible confounding factors that can affect the quality of sleep (age, biometric data, associated pathologies).

This study will require confirming the diagnosis of glaucoma in subjects declared as such, and specifying the stage of glaucomatous involvement. A current ophthalmologic examination of glaucoma assessment will therefore be offered to this group of subjects (including examination of the visual field and tomography of the optic nerve). This study will also require verifying with certainty the absence of glaucoma in subjects in the control group. To this end, a telephone questionnaire will be administered to the subjects of this group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in the MARS database of CHU Grenoble-Alpes with available polysomnographic data and with the following ophthalmological characteristics:
* Glaucoma group: increase in intraocular pressure (IOP before treatment greater than 21 mmHg) with characteristic alterations of the optic nerve (pathological papillary excavation, papillary pallor, papillary atrophy) with corresponding alterations and characteristics of the visual field. The visual field should be considered reliable (European criteria (European Glaucoma Society, 1999).
* Control group: no known ophthalmological pathologies, with an ophthalmological examination on telephone examination - in the 2 years preceding the polysomnographic examination - normal apart from minor refractive disorders (myopia with spherical equivalent less than -6 diopters or hyperopia with spherical equivalent less than 3 diopters).
* Patients whose age is greater than or equal to 18 years
* Male or female patients
* Non-opposition to the study
* Affiliation to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Adult person under tutorship or curatorship or unable to express their consent / opposition
* Person deprived of liberty
* Opposition expressed to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our population is taken from the MARS database. The MARS database (Multimorbidity Apnea Respiratory failure Sleep database) is a database designed by the EFCR CHU Grenoble Alpes laboratory.
  It consists of patients with respiratory pathology associated or not with other pathologies and patients with respiratory pathology associated with several co-morbidities.
  It is a database that has so far received all the legal authorizations required for its use and scientific exploitation (CCTIRS: Request for advice N ° 15.925bis, favorable opinion obtained on 03/23/2016; CNIL: Declaration of conformity to the reference methodology MR003 N ° 1996650v0 on 05/10/2016). This database is also managed in compliance with GDPR rules.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
To study the polysomnographic characteristics of sleep in glaucomatous and non-glaucomatous subjects | Baseline (PSG)
  Total sleep time in glaucomatous and control subjects

SECONDARY OUTCOMES:
To characterize of the architecture of sleep in glaucomatous and non-glaucomatous subjects. | Baseline (PSG)
  Length of sleep period Time spent in phase 1, 2, 3 and 4 Micro-alarm clocks index Time with saturation less than 90% Apnea-hypopnea index

IPD SHARING:
Plan to Share IPD: Undecided